CLINICAL TRIAL: NCT06708260
Title: A Phase 2, Multicenter, Randomized, Parallel Study to Evaluate the Efficacy and Safety of Two Doses of ENN0403 in Subjects with Diabetic Macular Edema (DME)
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of ENN0403 in Subjects with DME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EnnovaBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENN0403-P2-CN-03
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Macular Edema (DME)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ENN0403 low dose treatment arm (Experimental)
  Interventions: Drug: ENN0403, low dose
- ENN0403 high dose treatment arm (Experimental)
  Interventions: Drug: ENN0403, high dose

INTERVENTIONS:
Drug: ENN0403, low dose — ENN0403 capsules will be orally administered once a day for 12 weeks.
  Arms: ENN0403 low dose treatment arm
Drug: ENN0403, high dose — ENN0403 capsules will be orally administered once a day for 12 weeks.
  Arms: ENN0403 high dose treatment arm

SUMMARY:
This is a multicenter, randomized, parallel study to evaluate the efficacy and safety of two doses of ENN0403 in subjects with diabetic macular edema (DME). Approximately 60 subjects will be randomized to receive ENN0403 capsule orally once a day at the low dose or high dose with a 1:1 ratio. The study period consisted of up to 2 weeks of screening, 12 weeks of treatment and 2 weeks of follow-up, and the entire trial period was up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent;
2. Aware of the entire study process and requirements, understands the importance of medication compliance and completing all assessments on time throughout the study, and agrees to strictly follow the protocol and study procedures, including restrictions on drug combination during the study;
3. Diagnosis of type 1 or type 2 diabetes mellitus and HbA1c≤10.0% with regular use hypoglycemic drugs and stable glycemic control 1 month before screening (at the discretion of the investigator);
4. The decrease of BCVA is mainly caused byDiabetic Macular Edema in the study eye;
5. BCVA letter score of ≤ 73 (Snellen 20/40) and ≥ 24 (Snellen 20/320) at screening visit and at baseline. If both eyes meet the inclusion criteria, the study eye will be determined by the investigator from a medical perspective. ( If both eyes meet the inclusion criteria，the eye with poor baseline vision will be selected as the study eye; If the BCVA number is the same, choose the eye with the thicker CRT as the study eye) ；
6. Optical Coherence Tomography (OCT) foveal CRT at screening measuring ≥300 μm.

Exclusion Criteria:

1. Study eye with any eye disease or medical history other than DME that causes or may cause irreversible vision loss;
2. Study eye had glaucoma filtration surgery in the past or may have the surgery during the study;
3. Study eye had previously undergone vitreoretinal surgery;
4. Study eye received intraocular hormone drugs within 6 months prior to baseline or periocular or systemic hormone drugs within 3 months prior to baseline;
5. Any eye received intraocular injection of VEGF within 3 months prior to baseline;
6. History of idiopathic or autoimmune uveitis in any eye;
7. Uncontrolled glaucoma in any eye (defined as IOP ≥25 mmHg after treatment with anti-glaucoma drugs)
8. History of allergy to the investigational drug or any ingredient, or to any ingredient used during the treatment;
9. Use of any other investigational drug or device within 3 months or 5 half-lives prior to baseline (whichever is longer);
10. Other factors considered inappropriate for inclusion in this study at the discretion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Central Retinal Thickness (CRT) at week 12 | week 12

SECONDARY OUTCOMES:
Change from baseline in Best Corrected Visual Acuity (BCVA) at week 4, 8, and 12 | week 4, 8, 12
Change from baseline in CRT at week 4 and 8 | week 4, 8
Incidence of ocular and non-ocular TEAE and SAE | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China